CLINICAL TRIAL: NCT01815749
Title: Phase I Study of Cellular Immunotherapy Using Central Memory-Enriched T Cells Lentivirally Transduced to Express a CD19-Specific, CD28-Costimulatory Chimeric Receptor and a Truncated EGFR Following Peripheral Blood Stem Cell Transplantation for Patients With High-Risk Intermediate Grade B-Lineage Non-Hodgkin Lymphoma
Brief Title: Genetically Modified T-cell Infusion Following Peripheral Blood Stem Cell Transplant in Treating Patients With Recurrent or High-Risk Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12224; NCI-2013-00590 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P50CA107399 (NIH)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2024-10

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (genetically modified T cell infusion) (Experimental): Patients undergo mobilization for autologous stem cell collection with cytoreductive chemotherapy and filgrastim and/or plerixafor per current standard operating policies. Patients undergo myeloablative conditioning regimen per institutional standards beginning day -7 followed by hematopoietic stem cell transplantation on day 0. Patients receive CD19-CAR-specific/truncated EGFR lentiviral vector-transduced autologous T cells IV on day 2 or 3 (may be delayed up to day 45 if the patient is not yet eligible). Patients who experience disease progression and have not experienced DLTs at greater than or equal to 100 days post HSCT will be allowed to receive an optional second T cell infusion.
  Interventions: Biological: autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tcm-enriched T cells; Procedure: autologous hematopoietic stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tcm-enriched T cells — Given IV
  Other Names: CD19-CAR-specific/truncated EGFR lentiviral vector-transduced autologous T cells
Procedure: autologous hematopoietic stem cell transplantation — Undergo autologous hematopoietic stem cell transplantation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of genetically modified T-cells following peripheral blood stem cell transplant in treating patients with recurrent or high-risk non-Hodgkin lymphoma. Giving chemotherapy before a stem cell transplant helps stop the growth of cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Removing the T cells from the donor cells before transplant may stop this from happening. Giving an infusion of the donor's T cells (donor lymphocyte infusion) later may help the patient's immune system see any remaining cancer cells as not belonging in the patient's body and destroy them (called graft-versus-tumor effect)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and describe the full toxicity profile of cellular immunotherapy utilizing ex vivo expanded autologous central memory T cell (Tcm)-enriched T cells that are genetically modified using a self-inactivating (SIN) lentiviral vector to express a costimulatory cluster of differentiation (CD)19-specific chimeric antigen receptors (CAR) as well as a truncated human epidermal growth factor receptor (EGFR) (CD19R:CD28 zeta/EGFR tau +Tcm) (CD19-CAR-specific/truncated EGFR lentiviral vector-transduced autologous T cells) in conjunction with a standard myeloablative autologous hematopoietic stem cell transplant (HSCT) for patients with high-risk intermediate grade B-lineage non-Hodgkin lymphoma (e.g., diffuse large B-cell lymphoma [DLBCL], mantle cell lymphoma [MCL] or transformed non-Hodgkin lymphoma [NHL]).

II. To determine the maximum tolerated dose (MTD) based on dose limiting toxicities (DLTs).

SECONDARY OBJECTIVES:

I. To determine the tempo, magnitude, and duration of engraftment of the transferred T cell product as it relates to the number of cells infused.

II. To study the impact of this therapeutic intervention on the development of normal CD19+ B-cell precursors in the peripheral blood as a surrogate for the in vivo effector function of transferred autologous CD19R:CD28 zeta/EGFR tau +Tcm.

OUTLINE: This is a dose-escalation study of CD19-CAR-specific/truncated EGFR lentiviral vector-transduced autologous T cells. Patients undergo mobilization for autologous stem cell collection with cytoreductive chemotherapy and filgrastim and/or plerixafor per current standard operating policies. Patients undergo myeloablative conditioning regimen per institutional standards beginning day -7 followed by hematopoietic stem cell transplantation on day 0. Patients receive CD19-CAR-specific/truncated EGFR lentiviral vector-transduced autologous T cells IV on day 2 or 3 (may be delayed up to day 45 if the patient is not yet eligible). Patients who experience disease progression and have not experienced DLTs at greater than or equal to 100 days post HSCT will be allowed to receive an optional second T cell infusion.

After completion of study treatment, patients are followed up weekly for 1 month, monthly for 1 year, and then yearly for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Research participants enrolled are patients with an indication to be considered for HSCT, who are diagnosed with intermediate grade B-cell NHL (e.g., DLBCL, MCL or transformed NHL), and that have either recurrence/progression following prior therapy, or verification of high-risk disease in first remission
* Karnofsky performance status of >= 70% and a life expectancy >= 16 weeks at time of enrollment
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* City of Hope (COH) pathology review confirms that research participant's diagnostic material is consistent with the history of intermediate grade B-cell NHL (e.g., DLBCL, MCL or transformed NHL)
* Negative serum pregnancy test for women of childbearing potential
* Research participant has an indication to be considered for autologous stem cell transplantation
* All patients must have the ability to understand and the willingness to sign a written informed consent

ELIGIBILITY TO UNDERGO AUTOLOGOUS MYELOABLATIVE TRANSPLANTATION WITH HEMATOPOETIC PROGENITOR CELL (HPC)A RESCUE

* Research participant meets all standard clinical parameters for candidates of autologous transplant as described in the current COH Hematopoietic Cell Transplant Standard Operating Policies, Procedures and Protocols
* Patient Evaluation & Selection or Deferral for hematopoietic cell transplantation (HCT)
* Research participant is scheduled to receive a standard chemotherapy-based conditioning regimen, such as cyclophosphamide, carmustine, etoposide (CBV) or carmustine, etoposide, cytarabine, melphalan (BEAM)
* Research participant has a cryopreserved unselected HPCA product of at least 3 x 10^6/kg CD34+ cells
* Research participant does not have evidence of disease progression after salvage therapy

ELIGIBILITY CRITERIA AT TIME OF INFUSION OF GENETICALLY MODIFIED AUTOLOGOUS T CELLS

* Research participant has a released cryopreserved T cell product
* Research participant has undergone an autologous HPC(A) procedure
* Not requiring supplemental oxygen or mechanical ventilation, oxygen saturation of 90% or higher on room air
* Not requiring pressor support, not having symptomatic cardiac arrhythmias
* Lack of acute renal failure/requirement for dialysis, as evidenced by creatinine < 1.6 - Total bilirubin =< 5.0
* Research participant without clinically significant encephalopathy/new focal deficits
* No clinical evidence of uncontrolled active infections process

Exclusion Criteria:

* Research participants with any uncontrolled illness including ongoing or active infection; research participants with known active hepatitis B or C infection; research participants who are human immunodeficiency virus (HIV) seropositive based on testing performed within 4 weeks of enrollment; research participants with any signs of symptoms of active infection, positive blood cultures or radiological evidence of infections
* Research participants receiving any other investigational agents, or concurrent biological, chemotherapy or radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cetuximab
* Research participants with known brain metastases (central nervous system [CNS] involvement or parenchymal or leptomeningeal involvement)
* Research participants with presence of other malignancy or history of prior malignancy within 5 years of study entry; although patients treated with curative intent within 5 year are eligible; this exclusion rule does not apply to non-melanoma skin tumors and in-situ cervical cancer
* Failure of research participant to understand the basic elements of the protocol and/or the risks/benefits of participating in this phase I/II study; a legal guardian may substitute for the research participant
* History of allogeneic HSCT or prior autologous HSCT
* Any standard contraindications to myeloablative HSCT per standard of care practices at COH
* Dependence on corticosteroids
* Active autoimmune disease requiring systemic immunosuppressive therapy
* Research participants will be excluded, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10-08 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events attributed to Tcm adoptive transfer as reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 15 years
  Tables will be created to summarize all toxicities and side effects by dose, course, organ, and severity.
MTD of CD19-CAR-specific/truncated EGFR lentiviral vector-transduced autologous T cells based on dose limiting toxicities | Up to day 28
  Graded according to the NCI CTCAE version 4.0.

SECONDARY OUTCOMES:
Engraftment of the transferred T cell products | Up to 21 days
  Rates and associated 95% confidence limits will be estimated.
CD19+ B cell precursors in the peripheral blood as a surrogate for the in vivo effector function of transferred CD19-specific T cells | Up to 28 days
  Rates and associated 95% confidence limits will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Budde, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Wang X, Popplewell LL, Wagner JR, Naranjo A, Blanchard MS, Mott MR, Norris AP, Wong CW, Urak RZ, Chang WC, Khaled SK, Siddiqi T, Budde LE, Xu J, Chang B, Gidwaney N, Thomas SH, Cooper LJ, Riddell SR, Brown CE, Jensen MC, Forman SJ. Phase 1 studies of central memory-derived CD19 CAR T-cell therapy following autologous HSCT in patients with B-cell NHL. Blood. 2016 Jun 16;127(24):2980-90. doi: 10.1182/blood-2015-12-686725. Epub 2016 Apr 26. PMID 27118452